CLINICAL TRIAL: NCT07098754
Title: Comparative Analysis of Different Physiotherapy Interventions on Craniovertebral Angle in Individuals With Myofascial Pain Syndrome and Radiculopathy: a Randomized Controlled Trial
Brief Title: Comparing Physical Therapy Interventions on Craniovertebral Angle (CVA) in Cervical Myofascial Pain Syndrome (MPS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Orthopedic and General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NOGH/NasirMehmoodPhD/0125/001
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Myofascial Pain Syndrome - Neck
Keywords: myofascial pain syndrome; dry needling in myofascial pain syndrome; cupping therapy in myofascial pain syndrome; best intervention for myofascial pain syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling; Transcutaneous Electric Nerve Stimulation; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dry Needling (Experimental): this group will receive dry needling with myofascial release
  Interventions: Other: Dry Needling
- Trigger Point Therapy (Experimental): this will receive trigger point therapy with stretching
  Interventions: Other: Trigger point therapy
- Cupping Therapy (Experimental): this will receive dry cupping therapy with Mobilizations Grade-1&2
  Interventions: Other: Maitlands' Mobilizations
- Conventional Physiotherapy (Active Comparator): Will receive electrotherapy with stretching and ROM exercises
  Interventions: Other: Tens and ultrasound

INTERVENTIONS:
Other: Dry Needling — will use dry needles of different recommended sizes to intercept the trigger points
  will add on myofascial release technique manually.
  Arms: Dry Needling
Other: Trigger point therapy — will release trigger points by manual pressure using trigger point therapy technique protocols
  will ad on stretching techniques
  Arms: Trigger Point Therapy
Other: Maitlands' Mobilizations — Maitlands' Mobilizations Grade-1& Grade-2 will be applied to upper thoracic and cervical regions
  dry cupping therapy will be applied as ad on therapy
  Arms: Cupping Therapy
Other: Tens and ultrasound — TENS and ultrasound will be applied according to recommended dosages followed by stretching and Range of motion activities
  Arms: Conventional Physiotherapy

SUMMARY:
Myofascial pain syndrome (MPS) and radiculopathy are prevalent musculoskeletal conditions that afflict a substantial portion of the population, causing significant discomfort and impairments in daily functioning. MPS is characterized by localized muscle pain, trigger points, and referred pain, often accompanied by stiffness and restricted range of motion. A common feature shared by individuals with MPS and radiculopathy is the presence of postural abnormalities and balance impairments . The craniovertebral angle, which reflects the relationship between the head and neck, is often compromised in these individuals due to muscle imbalances, pain-related guarding, and structural changes in the spine. Various physiotherapy modalities, including dry needling, manual mobilization and soft tissue release, trigger point therapy, stretching, cupping therapy, and electrotherapy, have been utilized in clinical practice, but their relative efficacy in improving the craniovertebral angle and alleviating symptoms in individuals with MPS and radiculopathy has not been comprehensively compared. Understanding the underlying mechanisms and comparative effectiveness of various physiotherapy interventions is essential for guiding evidence-based clinical decision-making and optimizing treatment outcomes for individuals with MPS and radiculopathy. By elucidating the effects of different treatment modalities on the craniovertebral angle and associated outcomes, this research endeavor aims to contribute to the development of more tailored and effective physiotherapy approaches for improving the well-being of individuals affected by these debilitating musculoskeletal conditions.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) and radiculopathy are prevalent musculoskeletal conditions that afflict a substantial portion of the population, causing significant discomfort and impairments in daily functioning. Myofascial pain syndrome (MPS) is characterized by localized muscle pain, trigger points, and referred pain, often accompanied by stiffness and restricted range of motion. Radiculopathy, on the other hand, involves dysfunction or compression of spinal nerve roots, resulting in symptoms such as radiating pain, numbness, and weakness along the affected nerve pathway. Both conditions can profoundly impact an individual's quality of life, leading to limitations in activities of daily living, work-related tasks, and recreational activities.

A common feature shared by individuals with Myofascial pain syndrome (MPS) and radiculopathy is the presence of postural abnormalities and balance impairments. The craniovertebral angle, which reflects the relationship between the head and neck, is often compromised in these individuals due to muscle imbalances, pain-related guarding, and structural changes in the spine. The alteration in the craniovertebral angle can exacerbate symptoms, contribute to muscle tension, and impede proper biomechanical function, further exacerbating the overall discomfort and functional limitations experienced by affected individuals.

The clinical examination of individuals with cervical spine disorders routinely encompasses assessment of posture, mobility, strength, and neuromuscular function. Among these, forward head posture (FHP)-characterized by anterior displacement of the head relative to the trunk-has been recognized as a key contributor to cervical dysfunction, neck pain, and related impairments. FHP is frequently implicated in a wide spectrum of musculoskeletal and neurological concerns, including temporomandibular disorders, headaches, visual disturbances, tinnitus, and altered electromyographic activity of craniofacial muscles, all of which can reduce sleep quality and daily function.

Anatomically, FHP involves extension of the upper cervical segments (C1-C3) and flexion of the lower cervical and upper thoracic segments, resulting in altered biomechanics and increased stress on the cervical musculature and joint. In addition, increased thoracic kyphosis is often associated with or predictive of FHP.

The craniovertebral angle (CVA), defined between a horizontal line through C7 and a line from C7 to the tragus of the ear, remains one of the most clinically accessible and valid quantitative indicators of FHP. A lower CVA represents a more pronounced forward head position, while higher angles reflect better postural alignment.

Despite these validated tools, there is limited research validating newer software platforms like MicroDiCom-commonly used in medical imaging-which may offer improved calibration, workflow integration, or measurement consistency. Each platform's unique interface and processing methodology necessitate separate psychometric evaluation.

Various physiotherapy modalities, including dry needling, manual mobilization and soft tissue release, trigger point therapy, stretching, cupping therapy, and electrotherapy, have been utilized in clinical practice, but their relative efficacy in improving the craniovertebral angle and alleviating symptoms in individuals with Myofascial pain syndrome (MPS)and radiculopathy has not been comprehensively compared.

Myofascial pain syndrome is often diagnosed in neuro-Musculo-skeletal pain patients with active Myofascial Trigger Points (MTrPs). The literature proposes many myo-fascial trigger point therapy procedures. There is a lack of credible evidence about inter and intra-efficacy among various therapy methods. One high-quality and two low-quality studies showed that conventional ultrasonography does not cure cervical and upper back myofascial trigger point pain better than placebo or no treatment. Magnet therapy may be a beneficial treatment, but more high-quality research is needed. Manual therapy trials imply that these therapies can be useful, however medium to long-term efficacy or effect more than placebo cannot be determined. Many neck region myofascial trigger point pain therapies lack proof. The variability of the included studies suggests that future high-quality trials could impact this review's conclusions. Future research must also examine perpetuating and contributory factors and the clinical efficacy of various treatment strategies.

Therefore, this research study aims to conduct a comparative analysis of these physiotherapy treatments on the craniovertebral angle in individuals diagnosed with MPS and radiculopathy. By evaluating the effects of different treatment modalities on posture, balance, pain levels, and overall quality of life, this study seeks to provide valuable insights into the optimal management of these challenging conditions.

Understanding the underlying mechanisms and comparative effectiveness of various physiotherapy interventions is essential for guiding evidence-based clinical decision-making and optimizing treatment outcomes for individuals with MPS and radiculopathy. By elucidating the effects of different treatment modalities on the craniovertebral angle and associated outcomes, this research endeavor aims to contribute to the development of more tailored and effective physiotherapy approaches for improving the well-being of individuals affected by these debilitating musculoskeletal conditions.

while there is evidence supporting the use of various physiotherapy interventions for managing pain and improving function in individuals with Myofascial pain syndrome (MPS) and radiculopathy, there is a paucity of research specifically comparative analysis of these interventions to find the most effective one as well as evaluating their effects on the craniovertebral angle. Addressing this gap in the literature is essential for developing more targeted and effective treatment approaches tailored to the unique needs of individuals with these conditions. The present study aims to fill this gap by conducting a comparative analysis of different physiotherapy treatments and their effects on the craniovertebral angle, pain levels, functional ability, and quality of life in individuals with MPS and radiculopathy.

Rationale:

Myofascial pain syndrome (MPS) and radiculopathy present complex challenges in clinical management, causing localized muscle pain, trigger points, and neurological deficits. These conditions severely impact daily functioning and quality of life, often manifesting in postural abnormalities and balance impairments. The craniovertebral angle, reflecting head-neck relationship, is frequently affected, leading to increased muscle tension and reduced mobility. Physiotherapy is pivotal in managing these conditions, yet the optimal approach targeting the craniovertebral angle remains unclear due to insufficient research. This study aims to compare various physiotherapy treatments (e.g., dry needling, manual mobilization) to improve the craniovertebral angle and alleviate symptoms. By understanding treatment effectiveness, healthcare providers can tailor interventions, ultimately improving care for MPS and radiculopathy patients. This research seeks to elucidate treatment mechanisms, guide clinical decisions, and enhance overall well-being for this challenging patient population

OBJECTIVES OF THE STUDY

Principal Objective:

To assess and compare the effects of different physiotherapy modalities, including dry needling, manual mobilization and soft tissue release, trigger point therapy, stretching, cupping therapy, and electrotherapy, on the craniovertebral angle and quality of life in individuals diagnosed with myofascial pain syndrome (MPS) and radiculopathy.

Specific Objectives:

1. To compare improvements in pain levels, functional ability, and overall quality of life among the different treatment groups.
2. To evaluate effects of different physiotherapy interventions on range of motion.
3. To evaluate the effects of different physiotherapy interventions on craniovertebral angle.
4. To evaluate the effects of different physiotherapy interventions on balance.
5. To evaluate effects of different physiotherapy interventions on quality of life.
6. To evaluate effects of different physiotherapy interventions on myofascial trigger points.

Research Question:

I. Which is the most effective physiotherapy intervention to treat abnormal craniovertebral angle in patients with myofascial pain syndrome (MPS) and radiculopathy? II. Which physiotherapy intervention can bring optimal improvements in pain levels, functional ability, and overall quality of life among patients with myofascial pain syndrome (MPS) and radiculopathy? III. What is the effectiveness of different physiotherapy interventions regarding pain in patients with myofascial pain syndrome (MPS) and radiculopathy? IV. What is the effectiveness of different physiotherapy interventions in improving craniovertebral angle in patients with myofascial pain syndrome (MPS) and radiculopathy? V. What is the effectiveness of different physiotherapy interventions in improving balance in patients with myofascial pain syndrome (MPS) and radiculopathy? VI. What is the effectiveness of different physiotherapy interventions for improving range of motion in patients with myofascial pain syndrome (MPS) and radiculopathy? VII. What are the effects of different physiotherapy interventions on quality of life among patients with myofascial pain syndrome (MPS) and radiculopathy?

Conceptual Framework of Study:

With the purpose of evaluating and contrasting the effects of various physiotherapy techniques on persons who have been diagnosed with myofascial pain syndrome (MPS) and cervical radiculopathy, this research study aims to conduct an investigation. This study will include a total of one hundred participants, and it will be divided into four unique treatment groups, which are as follows: In Group A, dry needling and myofascial release will be administered, in Group B, trigger point therapy and stretching will be performed, in Group C, mobilisation grade-1 and grade-2 will be performed in conjunction with cupping therapy, and in Group D, the control group, electrotherapy (TENS and ultrasound) will be administered in conjunction with stretching and range of motion exercises. It is the primary purpose of this study to assess the efficacy of the various physiotherapy methods with regard to the craniovertebral angle (CVA) and the overall quality of life. One of the specific goals is to evaluate the effects of the therapies on range of motion, balance, and myofascial trigger points. Other specific objectives include comparing the levels of pain, functional ability, and quality of life that have improved among the treatment groups. The various physiotherapy techniques that were utilized in this investigation are the independent factors. The dependent variables, on the other hand, consist of pain levels, functional capacity, quality of life, range of motion, craniovertebral angle, balance, and the existence of myofascial trigger points. A randomized controlled trial methodology will be utilized for the research project. This methodology will comprise the utilization of pre-, mid-, and post-intervention assessments to evaluate the dependent variables. Additionally, proper statistical analysis will be utilized to compare the outcomes across the different groups. In the end, the purpose of this research is to provide valuable insights into the effectiveness of various physiotherapy modalities for the management of myofascial pain syndrome and cervical radiculopathy, as well as their effects on the craniovertebral angle (CVA). These findings have the potential to guide clinical practice and improve patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Participants must be between 20 and 40 years old.
2. Gender: Both genders, Male and Female have equal chance of selection as participant in the study.
3. Diagnosis: Participants must have a confirmed diagnosis of myofascial pain syndrome (MPS), altered cervical posture, restricted range of motion of cervical spine due to muscular spasm etc, altered craniovertebral angle, pain in cervical region or upper extremity and/or radiculopathy by a qualified healthcare professional, based on standardized diagnostic criteria (e.g., clinical examination, imaging studies).
4. Severity: Participants should have mild to moderate symptoms of MPS and/or radiculopathy, as determined by the assessing healthcare provider.
5. Willingness to Participate: Participants must be willing and able to comply physically and mentally with the study procedures, including attending scheduled physiotherapy sessions and completing outcome assessments.
6. Informed Consent: Participants will have to provide written informed consent mendatorily to be selected as participant in the study after receiving detailed information about the study aims, procedures, potential risks, and benefits.

Exclusion Criteria:

1. Severe Comorbidities: Participants with severe comorbidities or medical conditions that may interfere with their ability to participate in the study or confound the interpretation of results will be excluded. C1, C2 compression… vertigo
2. Surgeries: Participants who have undergone surgeries in the cervical or head region in past will be excluded due to potential confounding effects on outcomes.
3. Pregnancy: Pregnant individuals will be excluded from the study due to the potential risks associated with certain physiotherapy modalities and the need for specialized considerations in this population.
4. Contraindications: Participants with contraindications to specific physiotherapy modalities included in the study protocol (e.g., contraindications to dry needling, electrotherapy) will be excluded to ensure participant safety.
5. Inability to Attend Sessions: Participants who are unable to attend scheduled physiotherapy sessions due to logistical constraints (e.g., transportation issues, scheduling conflicts) will be excluded.
6. Cognitive Impairment: Participants with significant cognitive impairment or communication difficulties that may impede their ability to understand and follow study instructions will be excluded.
7. Participation in Other Research: Participants who are currently participating in other research studies involving treatment interventions for MPS and/or radiculopathy will be excluded to avoid potential confounding effects on outcomes and treatment adherence.
8. Malignancies: participants suffering from any kind of malignancies will be excluded from the study.
9. Trauma: Participants having a history of trauma and fractures in head and neck region will also be excluded from the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral (CV) Angle | Four Weeks
  Angle between horizontal line crossing spinous process of C7 and line joining the same with tragus of ear.
  it is assessed using digital photography and then calculating angle using MicroDiCom Software.
Pain Severity | Four weeks
  Pain severity will be checked by Numeric Pain Rating Scale (NPRS). this scale consists of 0-10 values with 0 being no pain and 10 being the worst possible pain. Increasing pain scores show high severity of pain and decreasing/less scores show less severity of pain.

SECONDARY OUTCOMES:
Balance | Four weeks
  Balance will be assessed using Y Balance Test. this test measures distance of reach on posterior side, anterolateral and anteromedial sides of one leg from keeping one foot stationary on a center point. Distance/reach is measured in cm. Higher values show better balance then lower values of reach in any direction.

CONTACTS AND LOCATIONS:
Overall Officials: Mazhar A Professor, PhD, Study Chair — Nazeer Hussain University
Locations (1):
- National Orthopedic and General Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared due to ethical and confidentiality concerns

REFERENCES:
- [Result] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883
- [Result] Cheung Lau HM, Wing Chiu TT, Lam TH. Clinical measurement of craniovertebral angle by electronic head posture instrument: a test of reliability and validity. Man Ther. 2009 Aug;14(4):363-8. doi: 10.1016/j.math.2008.05.004. Epub 2008 Aug 9. PMID 18694655
- [Result] Al Bedah AM, Khalil MK, Posadzki P, Sohaibani I, Aboushanab TS, AlQaed M, Ali GI. Evaluation of Wet Cupping Therapy: Systematic Review of Randomized Clinical Trials. J Altern Complement Med. 2016 Oct;22(10):768-777. doi: 10.1089/acm.2016.0193. Epub 2016 Aug 24. PMID 27557333
- [Result] Joghataei MT, Arab AM, Khaksar H. The effect of cervical traction combined with conventional therapy on grip strength on patients with cervical radiculopathy. Clin Rehabil. 2004 Dec;18(8):879-87. doi: 10.1191/0269215504cr828oa. PMID 15609843
- [Result] Alfawaz S, Lohman E, Alameri M, Daher N, Jaber H. Effect of adding stretching to standardized procedures on cervical range of motion, pain, and disability in patients with non-specific mechanical neck pain: A randomized clinical trial. J Bodyw Mov Ther. 2020 Jul;24(3):50-58. doi: 10.1016/j.jbmt.2020.02.020. Epub 2020 Feb 22. PMID 32826008
- [Result] Mahajan R, Kataria C, Bansal K (2012). Comparative Effectiveness of Muscle Energy Technique and Static Stretching for Treatment of Subacute Mechanical Neck Pain. International Journal of Health and Rehabilitation Sciences; 1(1): 16-24.
- [Result] Arjona Retamal JJ, Fernandez Seijo A, Torres Cintas JD, de-la-Llave-Rincon AI, Caballero Bragado A. Effects of Instrumental, Manipulative and Soft Tissue Approaches for the Suboccipital Region in Subjects with Chronic Mechanical Neck Pain. A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Aug 16;18(16):8636. doi: 10.3390/ijerph18168636. PMID 34444389
- [Result] Wang SQ, Jiang AY, Gao Q. Effect of manual soft tissue therapy on the pain in patients with chronic neck pain: A systematic review and meta-analysis. Complement Ther Clin Pract. 2022 Nov;49:101619. doi: 10.1016/j.ctcp.2022.101619. Epub 2022 Jun 12. PMID 35988324
- [Result] Kalichman L, Ben David C. Effect of self-myofascial release on myofascial pain, muscle flexibility, and strength: A narrative review. J Bodyw Mov Ther. 2017 Apr;21(2):446-451. doi: 10.1016/j.jbmt.2016.11.006. Epub 2016 Nov 14. PMID 28532889
- [Result] Ümit Dündar, Özlem Solak, Fatma aml, Vural Kavuncu. (2010). Effectiveness of Ultrasound Therapy in Cervical Myofascial Pain Syndrome: A Double Blind, Placebo-Controlled Study. Turk J Rheumatol; 25: 110-5
- [Result] Siddique MAE, Rahman MM, Islam MS, Islam MW, Islam N, Uddin Z, et al. Physiotherapy versus pain medication for managing chronic Cervical Radiculopathy: protocol for a multi-arm parallel-group randomized clinical trial. F1000Research. 2023; 12:465.
- [Result] Titcomb DA, Melton BF, Miyashita T, Bland HW. The Effects of Postural Education or Corrective Exercise on the Craniovertebral Angle in Young Adults with Forward Head Posture: A Randomized Controlled Trial. Int J Exerc Sci. 2023 Aug 1;16(1):954-973. doi: 10.70252/PYPQ8483. eCollection 2023. PMID 37649869
- [Result] Amjad F, Mohseni-Bandpei MA, Gilani SA, Ahmad A, Hanif A. Effects of non-surgical decompression therapy in addition to routine physical therapy on pain, range of motion, endurance, functional disability and quality of life versus routine physical therapy alone in patients with lumbar radiculopathy; a randomized controlled trial. BMC Musculoskelet Disord. 2022 Mar 16;23(1):255. doi: 10.1186/s12891-022-05196-x. PMID 35296293
- [Result] Han SC, Harrison P. Myofascial pain syndrome and trigger-point management. Reg Anesth. 1997 Jan-Feb;22(1):89-101. doi: 10.1016/s1098-7339(06)80062-3. PMID 9010953
- [Result] Cao QW, Peng BG, Wang L, Huang YQ, Jia DL, Jiang H, Lv Y, Liu XG, Liu RG, Li Y, Song T, Shen W, Yu LZ, Zheng YJ, Liu YQ, Huang D. Expert consensus on the diagnosis and treatment of myofascial pain syndrome. World J Clin Cases. 2021 Mar 26;9(9):2077-2089. doi: 10.12998/wjcc.v9.i9.2077. PMID 33850927
- [Result] Galasso A, Urits I, An D, Nguyen D, Borchart M, Yazdi C, Manchikanti L, Kaye RJ, Kaye AD, Mancuso KF, Viswanath O. A Comprehensive Review of the Treatment and Management of Myofascial Pain Syndrome. Curr Pain Headache Rep. 2020 Jun 27;24(8):43. doi: 10.1007/s11916-020-00877-5. PMID 32594264

DOCUMENTS (3):
  • Study Protocol (2025-03-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT07098754/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT07098754/SAP_001.pdf
  • Informed Consent Form (2025-03-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT07098754/ICF_002.pdf